CLINICAL TRIAL: NCT02642419
Title: Atrial Fibrillation and Ischemic Events With Rivaroxaban in Patients With Stable Coronary Artery Disease Study (AFIRE Study)
Brief Title: Atrial Fibrillation and Ischemic Events With Rivaroxaban in Patients With Stable Coronary Artery Disease Study
Acronym: AFIRE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Japan Cardiovascular Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFIRE Study
Record Dates: First submitted 2015-10-21; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Rivaroxaban; Platelet Aggregation Inhibitors; Aspirin; Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental)
  Interventions: Drug: Rivaroxaban
- Rivaroxaban and single antiplatelet drug (Experimental)
  Interventions: Drug: Rivaroxaban and single antiplatelet drug (aspirin, clopidogrel or prasugrel)

INTERVENTIONS:
Drug: Rivaroxaban and single antiplatelet drug (aspirin, clopidogrel or prasugrel) — * Rivaroxaban will be orally administered after a meal at a dose of 15 mg if the creatinine clearance (CLcr) is 50 mL/min or more and at a dose of 10 mg if the CLcr is 15-49 mL/min (regardless of time)
  * Antiplatelet will be selected from aspirin or thienopyridine derivatives (clopidogrel or prasugrel)
    * Aspirin will be orally administered once a day at a dose of 81 mg or 100 mg
    * Clopidogrel will be orally administered once a day after a meal at a dose of 75 mg. The dose will be reduced to 50mg once a day depending on age, body weight or clinical findings.
    * Prasugrel will be orally administered once a day at a dose of 3.75 mg. If the body weight is 50kg or less a reduced dose(2.5 mg once a day) will be considered depending on the age, renal function or other bleeding and thrombotic risk.
  Arms: Rivaroxaban and single antiplatelet drug
Drug: Rivaroxaban — Rivaroxaban will be orally administered at a dose of 15 mg if the creatinine clearance (CLcr) is 50 mL/min or more and at a dose of 10 mg if the CLcr is 15-49 mL/min.
  Arms: Rivaroxaban

SUMMARY:
In patients with atrial fibrillation (AF) complicated with coronary artery disease (CAD), antiplatelet drugs are commonly used for the prevention of recurrence of stent thrombosis and cardiovascular events in combination with anticoagulant drugs. Based on the observations that the incidence of hemorrhagic complications increased when an antiplatelet drug was administered in combination with vitamin K antagonist (VKA), the guidelines for antithrombotic therapy after PCI in the US and EU recommend that DAPT (dual anti-platelets therapy) should be used in AF-complicated CAD patients for as short a time as possible following single anti-platelet and VKA, and that monotherapy with VKA should be started from one year after PCI. In 2013 the European Heart Rhythm Association (EHRA) published the guidelines for the use of NOACs in NVAF patients, which state that NOACs may have advantage to VKAs in terms of anti-thrombotic effects in NVAF patients undergoing PCI. However, no clinical evidence has ever been generated to reveal the efficacy and safety of mono-drug therapy with a NOACs in stable CAD patients one year or more after PCI.

AFIRE study is planned to evaluate the efficacy and safety of mono-drug therapy with a rivaroxaban in stable CAD patients. Among NOACs, rivaroxaban was chosen because of the evidence in Japanese patients and the results of a sub-analysis of ROCKET AF suggesting that rivaroxaban is more effective than VKA in reducing the incidence of myocardial infarction (MI).

DETAILED DESCRIPTION:
Study Design:prospective, randomized, open-label trial

Allocation:ratio to rivaroxaban monotherapy and rivaroxaban in co-administration with a single anti-platelet therapy is 1: 1 using WEB system

ELIGIBILITY:
Inclusion Criteria:

Patients with non-valvular atrial fibrillation complicated with stable coronary artery disease who are 20 years or older, with CHADS2 score are ≧1 , and that fulfill one of the following criteria and can provide written consent for participation in the present study will be eligible.

1. Patients who underwent percutaneous coronary intervention(PCI), including plain old balloon angioplasty(POBA), at least one year ago
2. Patients who have coronary stenosis requiring no percutaneous coronary intervention (50% or more stenosis) as indicated by coronary CT or coronary angiography(CAG)
3. Patients who underwent coronary artery bypass graft (CABG) at least one year ago

Exclusion Criteria:

* Patients for whom rivaroxaban is contraindicated
* Patients for whom aspirin, thienopyridine derivatives (clopidogrel or prasugrel) are contraindicated
* Patients who underwent PCI, including POBA, in the past one year
* Patients who are going to undergo revascularization
* Patients who have a past history of stent thrombosis
* Those who are going to undergo invasive surgery (excluding digestive endoscopy and biopsy)
* Patients who have active tumors
* Patients who have poorly-controlled hypertension (systolic blood pressure at hospital admission: 160 mmHg or more)
* Patients who cannot discontinue treatment with antiplatelet drugs (the physician in charge will make a decision on the basis of the lesion shape, lesion site and type of stents.)
* Patients judged as inappropriate for this study by investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of cardiovascular events | mean duration: 2 years, maximum duration: 3 years
  stroke, non-CNS embolism, myocardial infarction, unstable angina pectoris requiring revascularizations or all-cause mortality
Major bleeding defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria | mean duration: 2 years, maximum duration: 3 years

SECONDARY OUTCOMES:
Net adverse clinical and cerebral events (NACCE) | mean duration: 2 years, maximum duration: 3 years
  composite of all-cause death, myocardial infarction, stroke and major bleeding.
Ischemic cardiovascular events and death | mean duration: 2 years, maximum duration: 3 years
  * All-cause mortality
  * Cardiovascular death
  * non-cardiovascular death
  * Myocardial infarction
  * Unstable angina pectoris requiring revascularization
  * Ischemic stroke
  * Transient ischemic attack
  * non-CNS embolism (systemic embolism pulmonary embolism, deep vein thrombosis)
  * PCI/CABG
  * Stent thrombosis
  * Ischemic stroke and systemic embolism
All bleeding events | mean duration: 2 years, maximum duration: 3 years
Adverse events excluding hemorrhagic events | mean duration: 2 years, maximum duration: 3 years
Comparison of the primary endpoints, ischemic cardiovascular events and mortality between patients treated with aspirin and patients treated with thienopyridine derivatives | mean duration: 2 years, maximum duration: 3 years
Subgroup analysis of primary endpoints, ischemic cardiovascular events and mortality according to the CHADS2 score and CHA2DS2-VASc score | mean duration: 2 years, maximum duration: 3 years
Subgroup analysis of primary endpoints, ischemic cardiovascular events and mortality according to subject characteristics | mean duration: 2 years, maximum duration: 3 years
Subgroup analysis of major bleeding and all bleeding events according to the HAS-BLED score in patients with and without co-administration of antiplatelet drug and analysis of specificity and sensitivity | mean duration: 2 years, maximum duration: 3 years
Comparison of the incidence of bleeding events according to whether or not proton pump inhibitors (PPIs) are used | mean duration: 2 years, maximum duration: 3 years
Comparison of the incidence of the primary endpoints according to whether rivaroxaban is administered in the morning or evening | mean duration: 2 years, maximum duration: 3 years
  Primary endpoints include the composite endpoint of cardiovascular events (stroke, non-CNS embolism, myocardial infarction, unstable angina pectoris requiring revascularization or cardiovascular death) and major bleeding defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria.
Correlation of discontinuation of antithrombotic agents with ischemic cardiovascular events, bleeding events and adverse events | mean duration: 2 years, maximum duration: 3 years
Correlation of prothrombin time at trough with bleeding events and evaluation of the cutoff values in patients with and without co-administration of antiplatelet drug | mean duration: 2 years, maximum duration: 3 years
The incidence of the primary endpoints according to different rates of adherence | mean duration: 2 years, maximum duration: 3 years
  Primary endpoints include the composite endpoint of cardiovascular events (stroke, non-CNS embolism, myocardial infarction, unstable angina pectoris requiring revascularization or cardiovascular death) and major bleeding defined by the International Society on Thrombosis and Haemostasis (ISTH) criteria.
  The rate of adherence will be calculated by dividing the number of prescribed tablets by the period of treatment: e.g., if 240 tablets are prescribed for 300 days, the rate of adherence will be 80.0% (240/300).

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, Principal Investigator — Japan Cardiovascular Research Foundation
Locations (1):
- Japan Cardiovascular Research Foundation, Suita, Osaka, Japan

REFERENCES:
- [Derived] Yamaguchi J, Arashi H, Hagiwara N, Yasuda S, Kaikita K, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Matsui K, Ogawa H; AFIRE Investigators. Age-Stratified Effect of Rivaroxaban Monotherapy for Atrial Fibrillation in Stable Coronary Artery Disease: A Post Hoc Analysis of the AFIRE Randomized Clinical Trial. JAMA Cardiol. 2025 Aug 13;10(10):990-9. doi: 10.1001/jamacardio.2025.2611. Online ahead of print. PMID 40802193
- [Derived] Iijima R, Tokue M, Nakamura M, Yasuda S, Kaikita K, Akao M, Ako J, Matoba T, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H; AFIRE Investigators. Thrombocytopenia as a Bleeding Risk Factor in Atrial Fibrillation and Coronary Artery Disease: Insights From the AFIRE Study. J Am Heart Assoc. 2023 Oct 17;12(20):e031096. doi: 10.1161/JAHA.123.031096. Epub 2023 Oct 10. PMID 37815031
- [Derived] Ishii M, Kaikita K, Yasuda S, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Nishihara E, Nakamura S, Matsui K, Ogawa H, Tsujita K; AFIRE Investigators. Risk prediction score for clinical outcome in atrial fibrillation and stable coronary artery disease. Open Heart. 2023 May;10(1):e002292. doi: 10.1136/openhrt-2023-002292. PMID 37173099
- [Derived] Ishii M, Kaikita K, Yasuda S, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H, Tsujita K; AFIRE Investigators. Rivaroxaban Monotherapy in Atrial Fibrillation and Stable Coronary Artery Disease Across Body Mass Index Categories. JACC Asia. 2022 Aug 27;2(7):882-893. doi: 10.1016/j.jacasi.2022.08.004. eCollection 2022 Dec. PMID 36713761
- [Derived] Naito R, Miyauchi K, Yasuda S, Kaikita K, Akao M, Ako J, Matoba T, Nakamura M, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H; AFIRE Investigators. Rivaroxaban Monotherapy vs Combination Therapy With Antiplatelets on Total Thrombotic and Bleeding Events in Atrial Fibrillation With Stable Coronary Artery Disease: A Post Hoc Secondary Analysis of the AFIRE Trial. JAMA Cardiol. 2022 Aug 1;7(8):787-794. doi: 10.1001/jamacardio.2022.1561. PMID 35704345
- [Derived] Arashi H, Yamaguchi J, Hagiwara N, Yasuda S, Kaikita K, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Kimura K, Hirayama A, Matsui K, Ogawa H; AFIRE investigators. Rivaroxaban Underdose for Atrial Fibrillation with Stable Coronary Disease: The AFIRE Trial Findings. Thromb Haemost. 2022 Sep;122(9):1584-1593. doi: 10.1055/s-0042-1744543. Epub 2022 Jun 13. PMID 35697255
- [Derived] Matsui K, Yasuda S, Kaikita K, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Ogawa H. The impact of kidney function in patients on antithrombotic therapy: a post hoc subgroup analysis focusing on recurrent bleeding events from the AFIRE trial. BMC Med. 2022 Feb 25;20(1):69. doi: 10.1186/s12916-022-02268-6. PMID 35209924
- [Derived] Matoba T, Yasuda S, Kaikita K, Akao M, Ako J, Nakamura M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H; AFIRE Investigators. Rivaroxaban Monotherapy in Patients With Atrial Fibrillation After Coronary Stenting: Insights From the AFIRE Trial. JACC Cardiovasc Interv. 2021 Nov 8;14(21):2330-2340. doi: 10.1016/j.jcin.2021.07.045. PMID 34736731
- [Derived] Matsuzawa Y, Kimura K, Yasuda S, Kaikita K, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Hagiwara N, Hirayama A, Matsui K, Ogawa H; AFIRE Investigators. Antithrombotic Therapy for Atrial Fibrillation and Coronary Artery Disease in Patients With Prior Atherothrombotic Disease: A Post Hoc Analysis of the AFIRE Trial. J Am Heart Assoc. 2021 Nov 2;10(21):e020907. doi: 10.1161/JAHA.121.020907. Epub 2021 Oct 18. PMID 34658247
- [Derived] Kaikita K, Yasuda S, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H. Bleeding and Subsequent Cardiovascular Events and Death in Atrial Fibrillation With Stable Coronary Artery Disease: Insights From the AFIRE Trial. Circ Cardiovasc Interv. 2021 Nov;14(11):e010476. doi: 10.1161/CIRCINTERVENTIONS.120.010476. Epub 2021 Sep 3. PMID 34474583
- [Derived] Fukaya H, Ako J, Yasuda S, Kaikita K, Akao M, Matoba T, Nakamra M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H. Aspirin versus P2Y12 inhibitors with anticoagulation therapy for atrial fibrillation. Heart. 2021 Nov;107(21):1731-1738. doi: 10.1136/heartjnl-2021-319321. Epub 2021 Jul 14. PMID 34261738
- [Derived] Akao M, Yasuda S, Kaikita K, Ako J, Matoba T, Nakamura M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H. Rivaroxaban monotherapy versus combination therapy according to patient risk of stroke and bleeding in atrial fibrillation and stable coronary disease: AFIRE trial subanalysis. Am Heart J. 2021 Jun;236:59-68. doi: 10.1016/j.ahj.2021.02.021. Epub 2021 Feb 28. PMID 33657403
- [Derived] Yasuda S, Kaikita K, Akao M, Ako J, Matoba T, Nakamura M, Miyauchi K, Hagiwara N, Kimura K, Hirayama A, Matsui K, Ogawa H; AFIRE Investigators. Antithrombotic Therapy for Atrial Fibrillation with Stable Coronary Disease. N Engl J Med. 2019 Sep 19;381(12):1103-1113. doi: 10.1056/NEJMoa1904143. Epub 2019 Sep 2. PMID 31475793